CLINICAL TRIAL: NCT04208854
Title: Observational Study With Metronomic Oral Vinorelbine in Elderly Patients With Locally Advanced / Metastatic Non-small-cell Lung Cancer (NSCLC)
Acronym: VINORELBINA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Group of Endovascular Oncology (Other)
Collaborators: Azienda Sanitaria Ospedaliera (Other)
Responsible Party: Sponsor
Other Study IDs: VINORELBINA
Record Dates: First submitted 2019-12-20; First posted 2019-12-23 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Locally Advanced/ Metastatic NSCLC
MeSH Terms: interventions — Vinorelbine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VINORELBINA: Vinorelbine 40 mg (2 cps of 20 mg) three times a week (Monday. Wednesday, Friday), for the first 2 weeks.
  Starting from the third week, in the absence of any severe toxicity (≥ 3) and in the opinion of the clinician, the dosage can be increased to 50 mg (1 cps from 30 + 1 cps from 20 mg), three times a week ( Monday, Wednesday, Friday) continuously.
  The dosage of 40 or 50 mg is continued until progression, patient refusal or unacceptable toxicity (in the clinician's opinion).
  Interventions: Drug: Vinorelbine

INTERVENTIONS:
Drug: Vinorelbine — Vinorelbine 40 mg (2 cps of 20 mg) three times a week (Monday. Wednesday, Friday), for the first 2 weeks.
  Starting from the third week, in the absence of any severe toxicity (≥ 3) and in the opinion of the clinician, the dosage can be increased to 50 mg (1 cps from 30 + 1 cps from 20 mg), three times a week ( Monday, Wednesday, Friday) continuously.
  The dosage of 40 or 50 mg is continued until progression, patient refusal or unacceptable toxicity (in the clinician's opinion).

SUMMARY:
Vinorelbine is the first line reference drug in the elderly patient with locally advanced / metastatic non-small-cell lung cancer (NSCLC). The introduction of the oral formulation of vinorelbine has determined a further impulse to its use in 1st line and above all to its use as "metronomic" therapy. Metronomic chemotherapy offers the advantage of increasing the overall dosage of the drug administered, but reducing the side effects or making them more easily manageable; it is practically a question of administering fractionated doses of the drug continuously for long periods (generally up to the progression of unacceptable disease or toxicity). This study collects data on the efficacy and tolerability of oral metronomic vinorelbine in elderly patients with NSCLC, performed as per normal clinical practice.

DETAILED DESCRIPTION:
Vinorelbine is the first line reference drug in the elderly patient with locally advanced / metastatic non-small-cell lung cancer (NSCLC). The introduction of the oral formulation of vinorelbine has determined a further impulse to its use in 1st line and above all to its use as "metronomic" therapy. Metronomic chemotherapy offers the advantage of increasing the overall dosage of the drug administered, but reducing the side effects or making them more easily manageable; it is practically a question of administering fractionated doses of the drug continuously for long periods (generally up to the progression of unacceptable disease or toxicity). This study collects data on the efficacy and tolerability of oral metronomic vinorelbine in elderly patients with NSCLC, performed as per normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of histologically documented NSCLC (adenocarcinoma and squamous carcinoma), stage IIIB (not eligible for surgery or chemo-radiotherapy) and stage IV according to the 8th edition of TNM
* "Wild type" for EGFR, ALK and PDL-1
* Age ≥ 70 years
* PS 0 - 2
* Adequate medullary reserve (neutrophils> 1500; PLT> 100,000 mm3); hepatic / renal function preserved
* Written informed consent

Exclusion Criteria:

* Gastrointestinal disorders that contraindicate the intake of the capsules (type ulcerative colitis or Chron's disease).
* Performance Status ECOG ≥ 3

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: ELDERLY PATIENTS <70 YEARS OLD
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-04-18 (Estimated); Study Completion 2020-05-18 (Estimated)

PRIMARY OUTCOMES:
TUMOR RESPONSE | 6 MONTHS
  STABLE DISEASE
number of adverse events | 6 MONTHS
  TOLERANCE TO VINORELBINE

SECONDARY OUTCOMES:
PFS | 1 year
  PROGRESSION FREE SURVIVAL
OS | 1 YEAR
  OVERALLA SURVIVAL

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro, Yes, Italy

IPD SHARING:
Plan to Share IPD: No